CLINICAL TRIAL: NCT06876298
Title: Role of Uromodulin in Management of Multiple Myloma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Usra Mohamed Farag, Usra Mohamed farrag Ahmed, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: multiple myloma
Record Dates: First submitted 2025-03-02; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myloma
Keywords: uromodulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients that newly diagnosed multiple myeloma with and without renal impairment (Other): Measurement of serum uromodulin in patients that newly diagnosed multiple myeloma with and without renal impairment and follow up these patients for 1 year.
  * All patients will be included within certain inclusion criteria after written consent will be subjected to;
  * Full medical history and clinical examination
  * Imaging:
    * abdominal ultrasound.
    * bone scan or low dose CT for lytic lesions.
  * Laboratory tests:
    * complete blood count with blood film
    * serum creatinine and urea and estimated GFR according to CKD-EPI
    * urine analysis
    * C-reactive protein (CRP)
    * serum calcium
    * serum total proteins and serum albumin
    * serum uric acid
    * 24 hours urinary protein.
    * Urine and\or protein electrophoresis with Immunofixation.
    * Serum Free light chains
    * Beta 2 microglobulin.
    * LDH
    * Serum Uromodulin level quantitative test by ELISA technique at day 0, day 21 of 1st cycle and at the end of 2nd cycle of bortezomib based protocol of chemotherapy.
  * Renal biopsy if indicated.
  Interventions: Diagnostic Test: - Serum Uromodulin level quantitative test by ELISA technique at day 0, day 21 of 1st cycle and at the end of 2nd cycle of bortezomib based protocol of chemotherapy.

INTERVENTIONS:
Diagnostic Test: - Serum Uromodulin level quantitative test by ELISA technique at day 0, day 21 of 1st cycle and at the end of 2nd cycle of bortezomib based protocol of chemotherapy. — - Serum Uromodulin level quantitative test by ELISA technique at day 0, day 21 of 1st cycle and at the end of 2nd cycle of bortezomib based protocol of chemotherapy.
  Other Names: • All patients will be included within certain inclusion criteria after written consent will be subjected to; • Full medical history and clinical examination • Imaging: - abdominal ultrasound. - bone

SUMMARY:
• To Evaluate the role of uromodulin level in early diagnosis of cast nephropathy and to detect its prognostic value in multiple myeloma patients

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignant plasma cell disorder . It is the second most common hematologic malignancy worldwide . It accounts for 15%-20% of all hematologic malignancies and has a 5-year survival rate of 60% .

About 31% of newly diagnosed MM patients presented with renal impairment and about 6% to 13% need dialysis , which significantly increases morbidity and mortality, and limits treatment strategies . Most common renal disease in MM is myeloma cast nephropathy that derived from secreted free light chains that combined with uromodulin to form cast which obstructs the distal tubules and presented with severe acute kidney injury . Renal biopsy is the only method to accurately diagnose myeloma cast nephropathy.

Uromodulin, also known as Tamm-Horsfall protein, is a kidney specific glycoprotein which is produced only by the epithelial cells lining the thick ascending limb (85%-90%) and early distal convoluted tubule (10%-15%), and is released to urine and blood . About 200 mg/day of uromodulin is normally excreted in urine . Recently, uromodulin being involved in many pathological processes as hypertension, urinary tract infections, nephrolithiasis, chronic and acute kidney disease.

Limited is known about role of uromodulin in management of myeloma. Measurement of serum uromodulin in patients that newly diagnosed multiple myeloma with and without renal impairment and follow up these patients for 1 year may provide a useful non-invasive predictor of cast nephropathy and may has a prognostic value in myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old that newly diagnosed with multiple myeloma according to 2024 updates in diagnosis of multiple myeloma (10) with and without renal impairment at nephrology and haematology unit of internal medicine department.

Exclusion Criteria:

* any patient have evidence of renal impairment due to any cause other than multiple myeloma as diabetic nephropathy, hypertensive nephropathy or lupus nephritis ... etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2027-03-25 (Estimated); Study Completion 2027-03-25 (Estimated)

PRIMARY OUTCOMES:
To assess the predictive value of serum uromodulin level in newly diagnosed patients with multiple myeloma with and without renal impairment as non-invasive marker for myeloma cast nephropathy.. | 1 year
  measurement of serum uromodulin level by ELISA technique in newly diagnosed patients with multiple myeloma with and without renal impairment at 3 times during course Bortizomib based chemotherapy to assess if serum uromodulin level is higher in patients with multiple myloma and renal impairment than in those without renal impairment and to detect the most accurate time to measure serum uromodulin during the treatment course.

SECONDARY OUTCOMES:
To detect correlation between serum uromodulin level and risk stratification, staging and prognosis of newly diagnosed patients with multiple myeloma. | 1 year
  To detect the correlation between serum uromodulin level and risk stratification, staging and prognosis of newly diagnosed patients with multiple myelom during follow up of these patients for 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Eygpt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Rajkumar SV. Multiple myeloma: 2024 update on diagnosis, risk-stratification, and management. Am J Hematol. 2024 Sep;99(9):1802-1824. doi: 10.1002/ajh.27422. Epub 2024 Jun 28. PMID 38943315
- [Background] Kipp A, Olinger E. What Does Uromodulin Do? Clin J Am Soc Nephrol. 2020 Dec 31;16(1):150-153. doi: 10.2215/CJN.06390420. Epub 2020 Aug 24. No abstract available. PMID 32839194
- [Background] Pruijm M, Ponte B, Ackermann D, Paccaud F, Guessous I, Ehret G, Pechere-Bertschi A, Vogt B, Mohaupt MG, Martin PY, Youhanna SC, Nagele N, Vollenweider P, Waeber G, Burnier M, Devuyst O, Bochud M. Associations of Urinary Uromodulin with Clinical Characteristics and Markers of Tubular Function in the General Population. Clin J Am Soc Nephrol. 2016 Jan 7;11(1):70-80. doi: 10.2215/CJN.04230415. Epub 2015 Dec 18. PMID 26683888
- [Background] LaFavers KA, Micanovic R, Sabo AR, Maghak LA, El-Achkar TM. Evolving Concepts in Uromodulin Biology, Physiology, and Its Role in Disease: a Tale of Two Forms. Hypertension. 2022 Nov;79(11):2409-2418. doi: 10.1161/HYPERTENSIONAHA.122.18567. Epub 2022 Aug 12. PMID 35959659
- [Background] Rusing LZ, Kozakowski N, Jeryczynski G, Vospernik L, Riedl J, Reiter T, Gisslinger H, Agis H, Krauth MT. Renal outcome in multiple myeloma patients with cast nephropathy: a retrospective analysis of potential predictive values on clinical and renal outcome. Hematology. 2024 Dec;29(1):2311600. doi: 10.1080/16078454.2024.2311600. Epub 2024 Feb 8. PMID 38329272
- [Background] Dimopoulos MA, Merlini G, Bridoux F, Leung N, Mikhael J, Harrison SJ, Kastritis E, Garderet L, Gozzetti A, van de Donk NWCJ, Weisel KC, Badros AZ, Beksac M, Hillengass J, Mohty M, Ho PJ, Ntanasis-Stathopoulos I, Mateos MV, Richardson P, Blade J, Moreau P, San-Miguel J, Munshi N, Rajkumar SV, Durie BGM, Ludwig H, Terpos E; International Myeloma Working Group. Management of multiple myeloma-related renal impairment: recommendations from the International Myeloma Working Group. Lancet Oncol. 2023 Jul;24(7):e293-e311. doi: 10.1016/S1470-2045(23)00223-1. PMID 37414019
- [Background] Fermand JP, Bridoux F, Dispenzieri A, Jaccard A, Kyle RA, Leung N, Merlini G. Monoclonal gammopathy of clinical significance: a novel concept with therapeutic implications. Blood. 2018 Oct 4;132(14):1478-1485. doi: 10.1182/blood-2018-04-839480. Epub 2018 Jul 16. PMID 30012636
- [Background] He J, Schmerold L, Van Rampelbergh R, Qiu L, Potluri R, Dasgupta A, Li L, Li Y, Hu P, Nemat S, Smugar SS, Zeltzer P, Appiani C, Li Q, Mehra M, Richarz U. Treatment Pattern and Outcomes in Newly Diagnosed Multiple Myeloma Patients Who Did Not Receive Autologous Stem Cell Transplantation: A Real-World Observational Study : Treatment pattern and outcomes in patients with multiple myeloma. Adv Ther. 2021 Jan;38(1):640-659. doi: 10.1007/s12325-020-01546-0. Epub 2020 Nov 19. PMID 33211297
- [Background] Sperling AS, Anderson KC. Facts and Hopes in Multiple Myeloma Immunotherapy. Clin Cancer Res. 2021 Aug 15;27(16):4468-4477. doi: 10.1158/1078-0432.CCR-20-3600. Epub 2021 Mar 26. PMID 33771856
- [Background] Rajkumar SV. Multiple myeloma: Every year a new standard? Hematol Oncol. 2019 Jun;37 Suppl 1(Suppl 1):62-65. doi: 10.1002/hon.2586. PMID 31187526